CLINICAL TRIAL: NCT00951301
Title: Mangosteen Effects on Inflammatory Markers in Atrial Fibrillation Trial
Brief Title: Evaluate Use of Mangosteen Juice Added to Usual Care in Reducing Risk of Recurrent Atrial Fibrillation
Acronym: MRI-AF
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Significantly lower accrual rate than anticipated, time constraints.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-007749
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mangosteen juice (Active Comparator): subjects randomized 1:1 to this arm will receive juice containing the mangosteen ingredient
  Interventions: Drug: mangosteen juice
- placebo juice (Placebo Comparator): subjects randomized 1:1 to this arm will receive specially prepared juice not containing mangosteen ingredient
  Interventions: Drug: placebo juice

INTERVENTIONS:
Drug: mangosteen juice — 6 ounces of juice containing mangosteen taken twice daily, AM and PM, for 6 months duration of study participation.
  Other Names: Xango juice
  Arms: mangosteen juice
Drug: placebo juice — 6 ounces of specially prepared juice not containing mangosteen taken twice daily, AM and PM, for 6 months duration of the study participation.
  Arms: placebo juice

SUMMARY:
This study is being done to see if the addition of mangosteen juice to standard medical care will reduce the risk of atrial fibrillation (AF) recurrence following direct current (DC) cardioversion. The study will also look at the effects the mangosteen juice may have on biomarkers of inflammation and endothelial cell dysfunction (the tissue lining the arteries does not function properly).

DETAILED DESCRIPTION:
Mangosteen Effects on Inflammatory Markers in Atrial Fibrillation Trial is a study designed to test the primary hypothesis that a dietary supplement (Mangosteen) containing anti-inflammatory and anti-oxidant properties may effect the measured levels of inflammatory biomarkers. Secondarily, this study will compare the attenuation of markers of endothelial cell dysfunction including endothelial progenitor cells (EPCs), clinical levels of anticoagulation (INR), digoxin, lipids, and glycosylated hemoglobin (Hgb A1c), quality of life measurements, AF recurrences, and associated levels of inflammatory markers with those experiencing recurrent AF between the mangosteen group and the placebo group.

This trial will randomize 250 patients presenting to the Mayo Clinic Cardioversion Unit over one year to two groups including a mangosteen supplemented group versus a control group with placebo juice. Patients will be enrolled who have a history of paroxysmal, persistent, or longstanding persistent atrial fibrillation and excluded if they have a history of recent surgery, myocardial infarction, infection, collagen vascular disease with active inflammation, or thyroid disease. Furthermore, patients already on corticosteroids will be excluded. Patients will be evaluated at enrollment and followed at 3 months and 6 months with repeat ECG, laboratory testing of inflammatory biomarkers and endothelial function, as well as quality of life questions.

The trial will track the effect of natural juices containing anti-inflammatory and anti-oxidant properties on inflammatory markers, endothelial progenitor cells, and quality of life. This trial will attempt to determine if any dietary supplement effects to inflammatory markers correlate with the rate of recurrent AF in each of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study must meet all of the following criteria:

  * Age >18 years
  * Documented atrial fibrillation with a clinically indicated cardioversion.
  * Anticoagulation with therapeutic INR or PTT as per Mayo Clinic cardioversion guidelines.
  * Provision of written informed consent.

Exclusion Criteria:

* Subjects will be excluded if any of the following conditions apply:

  * Presence of atrial fibrillation secondary to a reversible cause such as thyrotoxicosis or alcohol use
  * Myocardial infarction within 1 month, CABG or cardiac surgery including surgical maze or AF radiofrequency ablation within the past 3 months
  * Presence of an implanted pacemaker, atrial defibrillator, or ventricular defibrillator
  * History of bleeding diathesis or coagulopathy
  * Known atrial thrombus or contra-indication to cardioversion
  * Active infection or collagen vascular disease with active inflammation
  * Current use of corticosteroids
  * Gastrointestinal (GI) or genitourinary bleed within the past six months requiring transfusion
  * Concomitant medical illness (i.e., cancer, congestive heart failure) that may preclude protocol compliance, confound data interpretation or limit life-expectancy to less than one year
  * Known allergy to juice components
  * Inability or refusal to cooperate with study procedures
  * Unsuccessful cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that the addition of mangosteen juice as a dietary supplement may reduce the measured levels of inflammatory biomarkers interleukin 1, interleukin 6, C-reactive protein (CRP), and tumor necrosis factor alpha (TNF a) etc). | 6 months

SECONDARY OUTCOMES:
attenuation of markers of endothelial cell dysfunction including endothelial progenitor cell (EPCs). | 6 months
Clinical levels of anticoagulation (INR), digoxin, CBC, lipids, and glycosylated hemoglobin (Hgb A1c). | 6 months
Quality of life | 6 months
AF recurrence rates between the mangosteen group and the placebo group | 6 months
Associated levels of inflammatory markers with those experiencing recurrent AF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No